CLINICAL TRIAL: NCT04694807
Title: The Efficacy of Group Versus Individual Cognitive Behavioural Therapy for Complicated Grief Reactions in Old Age: A Randomized Non-inferiority Trial
Brief Title: Cognitive Behavioural Therapy for Complicated Grief Reactions in Old Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Utrecht University (Other); The Danish National Center for Grief (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35880
Record Dates: First submitted 2020-12-16; First posted 2021-01-05 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Bereavement; Prolonged Grief Disorder; Depression; Anxiety; Posttraumatic Stress Disorder
MeSH Terms: conditions — Prolonged Grief Disorder; Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Block randomization with a 1:1 allocation ratio to individually delivered versus group-based CBTgrief at the clinic in Copenhagen, and with a 1:2 allocation ratio to individually delivered versus group-based CBTgrief at the clinic in Odense. Randomization is conducted by an independent employee at the Danish National Center for Grief (DNCG). The allocation will take place after completion of baseline questionnaire (T1).
Masking Description: However, the investigator, therapists, and participants are masked in terms of not knowing which treatment the participants will be randomized to until after the completion of baseline assessment (T1).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-based Cognitive Behavioural Therapy (Experimental): A group delivered treatment format of CBTgrief (12 sessions).
  Interventions: Behavioral: Group-based Cognitive Behavioural Therapy for Complicated Grief Reactions
- Individually delivered Cognitive Behavioural Therapy (Active Comparator): An individual delivered treatment format of CBTgrief (12 sessions).
  Interventions: Behavioral: Individually delivered Cognitive Behavioural Therapy for Complicated Grief Reactions

INTERVENTIONS:
Behavioral: Group-based Cognitive Behavioural Therapy for Complicated Grief Reactions — CBTgrief is a transdiagnostic psychotherapeutic treatment for complicated grief reactions, i.e., symptoms of prolonged grief disorder as well as post-loss depression, anxiety, and posttraumatic stress. The treatment manual is developed by Professor Paul A. Boelen. CBTgrief includes methods such as psycho-education, homework, exposure, alteration of grief-related negative automatic thoughts, behavioural activation, and goal-oriented work. CBTgrief consists of 12 sessions with a session duration of 2.25 hours for the group format.
  Group-based CBTgrief will follow the same content and exercises for each session as individually delivered CBTgrief.
  Other Names: Group CBTgrief
  Arms: Group-based Cognitive Behavioural Therapy
Behavioral: Individually delivered Cognitive Behavioural Therapy for Complicated Grief Reactions — CBTgrief is a transdiagnostic psychotherapeutic treatment for complicated grief reactions, i.e., symptoms of prolonged grief disorder as well as post-loss depression, anxiety, and posttraumatic stress. The treatment manual is developed by Professor Paul A. Boelen. CBTgrief includes methods such as psycho-education, homework, exposure, alteration of grief-related negative automatic thoughts, behavioural activation, and goal-oriented work. CBTgrief consists of 12 sessions with a session duration of 1 hour for the individually delivered format.
  Individually delivered CBTgrief will follow the same content and exercises for each session as group-based CBTgrief.
  Other Names: Individual CBTgrief
  Arms: Individually delivered Cognitive Behavioural Therapy

SUMMARY:
While most bereaved individuals cope adaptively with the loss of a loved one, a significant minority experiences more severe and complicated grief reactions. Complicated grief reactions is an umbrella term for different types of post-loss complications, including symptoms of Prolonged Grief Disorder (PGD), depression, anxiety, and posttraumatic stress. These post-loss complications may all cause persistent suffering and functional impairment, thus pointing to a need for efficacious treatment.

While Cognitive Behavioural Therapy (CBT) is a relatively well-documented efficacious treatment for symptoms of PGD, depression, anxiety, and posttraumatic stress in the period after a loss, the relative efficacy of a transdiagnostic individually delivered versus group-based CBT for these types of complicated grief reactions (CBTgrief) remain unknown. Furthermore, little evidence exists about the relative cost-effectiveness of individually delivered versus group-based CBTgrief and why and how it works. The theory of CBTgrief proposes that it works by targeting three maintaining mechanisms in PGD: 1) Insufficient integration of the loss, 2) negative loss-related cognitions, and 3) depressive and anxious avoidance. These maintaining mechanisms have also shown to be statistically associated with depression, anxiety, and posttraumatic stress in the period after a loss, suggesting that different types of complicated grief reactions might share some of the same maintaining mechanisms. However, this proposed theory of change has yet to be empirically tested as a whole.

These knowledge gaps are crucial for the understanding of efficacious and cost-effective treatment formats as well as central treatment mechanisms in the psychological treatment of complicated grief reactions. The present study thus aims to examine the relative efficacy of an individually delivered versus group-based CBTgrief by means of a randomized non-inferiority trial. Secondary aims include an investigation of the relative cost-effectiveness of individually delivered versus group-based CBTgrief as well as treatment mediators. Finally, explorative analyses of potential moderators of intervention effects of CBTgrief will be conducted.

DETAILED DESCRIPTION:
Aims of the study:

1. Evaluate the relative efficacy of an individually delivered versus group-based CBTgrief.
2. Evaluate the relative cost-effectiveness of an individually delivered versus group-based CBTgrief.
3. Examine the theoretically proposed treatment mediators of CBTgrief.
4. Explore loss-related and sociodemographic characteristics as possible moderators of intervention effects.

Primary hypothesis:

Group-based CBTgrief will show non-inferiority (i.e., equal efficacy) in reducing symptoms of PGD compared to individually delivered CBTgrief at six months follow-up.

Secondary hypotheses:

1. Group-based CBTgrief will show non-inferiority (i.e., equal efficacy) in reducing symptoms of posttraumatic stress, depression, and anxiety compared to individually delivered CBTgrief at six months follow-up.
2. Group-based CBTgrief will be more cost-effective than individually delivered CBTgrief.
3. The observed effect of CBTgrief is mediated by changes in theoretically proposed maintaining mechanisms of complicated grief reactions (i.e. insufficient integration of the loss; negative loss-related cognitions; depressive and anxious avoidance).
4. Gender, level of education, age, baseline grief symptom level, type of loss, circumstances of the loss, time since loss, and number of additional losses will moderate the observed effects of CBTgrief.
5. Additional exploratory analyses include an additional matched comparison group, who have not received treatment in order to compare the effect of individual and group-based CBTgrief to a non-treatment group. This group will be extracted from a large-scale survey study: The Aarhus Bereavement Study (NCT03049007). Here, it is hypothesized that CBTgrief will have a statistically significant medium size effect on symptoms of PGD at six months follow-up compared to a matched comparison group, who did not receive treatment.

Design: The present study is conducted as a randomized non-inferiority trial of individually delivered versus group-based CBTgrief using block randomization.

Participants: Participants are recruited from the Danish National Center for Grief (DNCG), which is a Danish national organization that provide specialized psychological therapy to bereaved individuals who have lost a loved one. The therapists at the DNCG will screen and treat bereaved elderly people for complicated grief reactions with CBTgrief at their clinics in Odense and Copenhagen, Denmark. DNCG identifies participants through consultants, local practitioners, self-referral, and the DNCG grief support line.

Assessment points: Participants will be assessed at pre-, mid-, and post-intervention as well as at three and six months follow-up (T1-T5). Additionally, data on healthcare utilization will be retrieved from the Danish national registers concerning use of health care services such as visits to general practitioners, psychologists etc.

Sample size: A group sample size of 2x64 will enable us to detect non-inferiority between individually delivered and group-based CBTgrief with a non-inferiority of -0.5 SD on the primary outcome, i.e. symptoms of PGD, and a statistical power of 0.80. The true difference is assumed to be 0.0 and the one-sided significance level (alpha) of the test is 0.025. Based on an estimated dropout rate of 20% the total number of participants needed to recruit is N=160 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years (older adult).
2. Lost a loved one (e.g., spouse, partner) ≥ 6 months ago.
3. Clinically relevant symptoms of one or more types of complicated grief reactions (i.e. symptoms of prolonged grief (PG-13 ≥ 29), depression (CESD-10 ≥ 10), anxiety (GAD-7 ≥ 10), and/or posttraumatic stress (PCL ≥ 31)).

Exclusion Criteria:

1. No clinically relevant symptoms of one or more types of complicated grief reactions (i.e. symptoms of prolonged grief, depression, anxiety and/or posttraumatic stress).
2. No informed consent given.
3. Insufficient Danish proficiency.
4. Inability to transport oneself to the clinic.
5. Severe psychopathology (e.g., schizophrenia).
6. Severe cognitive impairment (e.g., Alzheimer's disease).
7. Substance abuse.
8. Acute suicidal ideation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 113 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Symptoms of prolonged grief disorder | From baseline (T1) to post-intervention (T3; up to one week after the 12th session) and to six months follow-up (T5).
  Changes in symptoms of prolonged grief disorder will be measured with Prolonged Grief Disorder-13 (PG-13; Prigerson et al., 2009). Higher total scores indicate higher symptom level (minimum value: 11; maximum value: 57).

SECONDARY OUTCOMES:
Depressive symptoms | From baseline (T1) to post-intervention (T3; up to one week after the 12th session), three months follow-up (T4), and six months follow-up (T5).
  Changes in depressive symptoms will be measured with Center for Epidemiologic Studies Short Depression Scale (CESD-10; Andresen, Malmgren, Carter, & Patrick, 1994). Higher total scores indicate higher symptom level (minimum value: 0; maximum value: 30).
Anxiety symptoms | From baseline (T1) to post-intervention (T3; up to one week after the 12th session), three months follow-up (T4), and six months follow-up (T5).
  Changes in anxiety symptoms will be measured with Generalized Anxiety Disorder-7 (GAD-7; Spitzer, Kroenke, Williams, & Löwe, 2006). Higher total scores indicate higher symptom level (minimum value: 0; maximum value: 21).
Posttraumatic stress symptoms | From baseline (T1) to post-intervention (T3; up to one week after the 12th session), three months follow-up (T4), and six months follow-up (T5).
  Changes in posttraumatic stress symptoms will be measured with Posttraumatic Stress Disorder Checklist for the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5) (PCL; Ashbaugh, Houle-Johnson, Herbert, El-Hage, & Brunet, 2016; Weathers et al., 2013). Higher total scores indicate higher symptom level (minimum value: 0; maximum value: 80).
Quality adjusted life years | From baseline (T1) to post-intervention (T3; up to one week after the 12th session), three months follow-up (T4), and six months follow-up (T5).
  Changes in quality adjusted life years will be assessed with 5Q-5D-5L (EuroQol Research Foundation, 2019) and used in order to evaluate cost-effectiveness.
Functional impairment | From baseline (T1) to post-intervention (T3; up to one week after the 12th session), three months follow-up (T4), and six months follow-up (T5).
  Changes in functional impairment will be measured with Sheehan Disability Scale (SDS; Leon, Olfson, Portera, Farber, & Sheehan, 1997). Higher total scores indicate greater functional impairment (minimum value: 0; maximum value: 30).
Loneliness | From baseline (T1) to post-intervention (T3; up to one week after the 12th session), three months follow-up (T4), and six months follow-up (T5).
  Changes in loneliness will be measured with Three-Item Loneliness Scale (TILS; Hughes, Waite, Hawkley, & Cacioppo, 2004). Higher total scores indicate greater loneliness (minimum value: 3; maximum value: 9).
Mental and physical function | From baseline (T1) to post-intervention (T3; up to one week after the 12th session), three months follow-up (T4), and six months follow-up (T5).
  Changes in mental and physical function will be measured with 12-Item Short Form Health Survey (SF-12; Ware, Kosinski, & Keller, 1996).
Social support | From baseline (T1) to post-intervention (T3; up to one week after the 12th session), three months follow-up (T4), and six months follow-up (T5).
  Changes in social support will be measured with Crisis Social Support scale (CSS; Joseph, Andrews, Williams, & Yule, 1992). Higher total scores indicate higher level of support (minimum value: 7; maximum value: 49).
Well-being | From baseline (T1) to post-intervention (T3; up to one week after the 12th session), three months follow-up (T4), and six months follow-up (T5).
  Changes in well-being will be measured with the five-item WHO Well-Being Index (WHO-5; Heun, Bonsignore, Barkow, & Jessen, 2001). Higher total scores indicate higher well-being (minimum value: 0; maximum value: 100).
Symptoms of prolonged grief disorder (at three months follow-up) | From baseline (T1) to three months follow-up (T3).
  Changes in symptoms of prolonged grief disorder will be measured with Prolonged Grief Disorder-13 (PG-13; Prigerson et al., 2009). Higher total scores indicate higher symptom level (minimum value: 11; maximum value: 57).
Symptoms of ICD-11 prolonged grief disorder | From baseline (T1) to post-intervention (T3; up to one week after the 12th session), three months follow-up (T4), and six months follow-up (T5).
  Changes in symptoms of ICD-11 prolonged grief disorder (i.e. the 11th revision of the International Classification of Diseases definition) will be measured by mapping questionnaire items from Prolonged Grief Disorder-13 (PG-13; Prigerson et al., 2009); Inventory of Complicated Grief Revised (ICG-r; Prigerson & Jacobs, 2001); Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5; Ashbaugh et al., 2016; Weathers et al., 2013).

OTHER OUTCOMES:
Mediator: Insufficient integration of the loss | Baseline (T1), mid-intervention (T2; immediately after the 6th session), post-intervention (T3; up to one week after the 12th session), three months follow-up (T4), six months follow-up (T5).
  Changes in the integration of the loss will be measured with Experienced Unrealness Scale (EUS; Boelen, 2010). Higher total scores indicate greater sense of unrealness (minimum value: 5; maximum value: 40).
Mediator: Negative loss-related cognitions | Baseline (T1), mid-intervention (T2; immediately after the 6th session), post-intervention (T3; up to one week after the 12th session), three months follow-up (T4), six months follow-up (T5).
  Changes in grief-related cognitions will be measured with Grief Cognitions Questionnaire (GCQ; Boelen & Lensvelt-Mulders, 2005). Higher total scores indicate higher levels of negative loss-related cognitions (minimum value: 0; maximum value: 90).
Mediator: Avoidance behaviors | Baseline (T1), mid-intervention (T2; immediately after the 6th session), post-intervention (T3; up to one week after the 12th session), three months follow-up (T4), six months follow-up (T5).
  Changes in avoidance behaviors will be measured with Depressive and Anxious Avoidance in Prolonged Grief Questionnaire (DAAPGQ; Boelen & van den Bout, 2010). Higher total scores indicate higher levels of avoidance behaviors (minimum value: 9; maximum value: 63).
Mediator: Therapeutic alliance | Mid-intervention (T2; immediately after the 6th session), post-intervention (T3; up to one week after the 12th session).
  Changes in the therapeutic alliance will be measured with Working Alliance Inventory - Short Form (WAI-SF; Horvath & Greenberg, 1989; Tracey & Kokotovic, 1989).
Mediator: Therapeutic group processes | Mid-intervention (T2; immediately after the 6th session), post-intervention (T3; up to one week after the 12th session).
  Changes in therapeutic group processes will be measured with Therapeutic Factors Inventory - Short Form (TFI-SF; Joyce, MacNair-Semands, Tasca, & Ogrodniczuk, 2011).
Healthcare utilization costs | Baseline (T1) to six months follow-up (T5).
  Data about visits to general practitioners, psychologists etc. delivered by the Danish Health Data Authority.
Moderator: Circumstances of the loss | Measured at baseline (T1).
  Data about circumstances of the loss (e.g., traumatic, non-traumatic) will be explored as a possible moderator.
Moderator: Type of loss | Measured at baseline (T1).
  Data about type of loss (e.g., spouse, child) will be explored as a possible moderator.
Moderator: Time since loss | Measured at baseline (T1).
  Data about time since loss will be explored as a possible moderator.
Moderator: Baseline grief symptom level | Measured at baseline (T1).
  Grief symptom level prior to intervention will be measured with Prolonged Grief Disorder-13 (PG-13; Prigerson et al., 2009) and explored as possible moderator.
Moderator: Number of additional losses | Measured at baseline (T1).
  Data about number of additional losses will be explored as a possible moderator.
Moderator: Sociodemographic characteristics (e.g., gender, age, level of education) | Measured at baseline (T1).
  Data about gender, age, level of education will be explored as possible moderators.

CONTACTS AND LOCATIONS:
Overall Officials: Maja O'Connor, PhD, Study Director — University of Aarhus
Locations (1):
- Unit for Bereavement Research, Dept. of Psychology, Aarhus University, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Komischke K, Boelen PA, Maccallum F, O'Connor M. Group Vs Individual Grief-Focused Cognitive Behavioral Therapy for Older Adults: A Randomized Clinical Trial. JAMA Psychiatry. 2026 Jan 14. doi: 10.1001/jamapsychiatry.2025.4106. Online ahead of print. PMID 41533372
- See also: Link to the research unit's website — https://psy.au.dk/en/research/research-centres-and-units/unit-for-bereavement-research/

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-07-04): https://cdn.clinicaltrials.gov/large-docs/07/NCT04694807/SAP_000.pdf